CLINICAL TRIAL: NCT05253976
Title: Post-market Clinical Follow-up Study to Confirm Safety, Performance and Clinical Benefits Data of the NexGen® Trabecular Metal™ (TM) Augmentation Patella (Implants and Instrumentation)- A Retrospective and Prospective Consecutive Series Study
Brief Title: PMCF Study on the Safety, Performance and Clinical Benefits Data of the NexGen TM Augmentation Patella
Status: Withdrawn | Type: Observational
Why Stopped: Study had to be terminated before first patient got enrolled due to insufficient case number.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-157K
Record Dates: First submitted 2022-01-12; First posted 2022-02-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2022-10

CONDITIONS: Rheumatoid Arthritis; Non-inflammatory Degenerative Joint Disease; Functional Deformity; Revision Total Knee Arthroplasty
Keywords: Post-Market Clinical Follow-Up Study; Medical Device; Performance; Safety; Clinical Benefits
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who received the NexGen TM Augmentation Patella

SUMMARY:
The study is a single-center, retrospective and prospective, non-randomized, non-controlled and consecutive series post-market study. The purpose of this study is to confirm safety, performance and clinical benefits of the NexGen TM Augmentation Patella. The primary objective is the assessment of safety by analyzing implant survivorship. This will be established by recording the incidence and frequency of revisions, complications and adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified.

The secondary objective is the assessment of performance and clinical benefits by recording patient-reported clinical outcome measures (PROMs) as well as radiographic outcomes.

DETAILED DESCRIPTION:
The Nexgen TM Augmentation Patella is intended to help compensate for significant bone loss in the patella during revision total knee arthroplasty.

One site will be involved in this study. The aim is to include a total of 25 consecutive series patients who received the NexGen TM Augmentation Patella starting from 2014 at the Inselspital Bern. All potential study subjects will be required to participate in the Informed Consent Process.

Baseline data from the preop, intraop and immediate post-op intervals will be available in medical notes and collected retrospectively. During follow-up visits at 1, 3, 5, 7 and 10 years post-op (depending on patients' date of surgery), the patient will be asked to complete patient questionnaires. Moreover, a clinical assessment and a radiographic evaluation will be conducted. In addition, any complications and adverse events will also be collected during these follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Non-inflammatory degenerative joint disease including osteoarthritis or traumatic arthritis
* Rheumatoid arthritis
* Correction of functional deformity
* Revision procedures where other treatments or devices have failed
* Treatment of fractures that are unmanageable using other techniques
* Complication from a failed prosthesis
* For cementless use only
* Supplemental fixation, when required, must be achieved by means of suture attachment.

Exclusion Criteria:

* Off-label use
* Primary arthroplasty
* Overt Infection
* Distant foci of infection (which may spread hematogenously to the implant site)
* Rapid disease progression as manifested by joint destruction or bone resorption apparent on roentgenogram
* Skeletally immature patients
* Cases where there is inadequate bone stock or no bone stock which would make the procedure unjustifiable
* Patients who are not willing to return for study required follow-up visits and/or are not willing to comply with the follow-up schedule
* Patient who is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, a known alcohol or drug abuser, anticipated to be non-compliant, younger than 18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of a consecutive series of patients who have been operated with the NexGen TM Augmentation Patella according to Zimmer Biomet's Instruction for Use (IFU) and who meet the inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and frequency of revisions, complications and adverse events. | From operation to study completion, 3-10 years
  Safety will be assessed by recording and analyzing the incidence and frequency of revisions, complications and adverse events.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | From post-operative to final follow-up visit, 3-10 years
  The KOOS assesses the patient's opinion about their knee and associated problems and consists of 5 subscales. Standardized answer options are given and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
EuroQol five-dimensional Health Questionnaire (EQ-5D-5L). | From post-operative to final follow-up visit, 3-10 years
  The EQ-5D-5L is a generic instrument . The EQ is scored on a 0 to 100 mm scale representing "the worst..." and "the best health you can imagine", respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (1):
- Insel Spital, Bern, Switzerland